CLINICAL TRIAL: NCT05396144
Title: Evaluation of Nitrous Oxide Use in GI Endoscopy Procedures: Potential for Optimizing Sedation and Minimizing Side-Effects During Recovery
Brief Title: Can Nitrous Oxide (Laughing Gas) be Used as a Sedative for GI Endoscopy Procedures?
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tim Angelotti, Associate Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 54961
Record Dates: First submitted 2022-05-12; First posted 2022-05-31 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Endoscopy; Colonoscopy
Keywords: sedative
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either receive 5% or 50% inhaled nitrous oxide in addition to typical sedative agents which will be given at the direction of the doctor performing the procedure. There is a 50% chance you will be assigned to receive either 5% or 50% nitrous oxide
Who Masked: Participant, Care Provider
Masking Description: The patient and healthcare providers (e.g. gastroenterologist performing the procedure and nurse administering conscious sedation) will not know if the patient is receiving either 5% or 50% inhaled nitrous oxide
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5% inhaled nitrous oxide (Sham Comparator): Patients will received 5% nitrous oxide by face mask in addition to standard intravenous sedatives given at the discretion of the care provider.
  Interventions: Drug: Nitrous oxide
- 50% inhaled nitrous oxide (Active Comparator): Patients will received 50% nitrous oxide by face mask in addition to standard intravenous sedatives given at the discretion of the care provider.
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Drug: Nitrous oxide — Nitrous oxide will be administered by face or nasal mask to be inhaled by the patient

SUMMARY:
Nitrous oxide (commonly known as 'laughing gas') is often used during dental and other outpatient procedures, because it is easy to administer, is short-acting and rapidly clears from the body following the procedure.

The investigators hypothesize that use of Nitrous oxide during GI endoscopy may enhance patient comfort during the procedure and speed-up post-procedure recovery, while minimizing the fatigue and mental fogginess some patients report the day after receiving standard sedative and narcotic drugs used routinely for the procedure.

The investigators are interested in determining if adding Nitrous Oxide to commonly used sedation drugs will decrease fatigue, mental fogginess, and nausea/vomiting, as well as determine when the patient felt fully recovered from the effects of all sedatives given for the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant patients age 18 and older
* Patient's presenting for upper endoscopy or colonoscopy under endoscopist- directed nurse sedation.
* Patient is willing and able to consent and comply with study procedures.

Exclusion Criteria:

* Age <18
* Potentially vulnerable subjects including, homeless people, pregnant females, employees and students.
* Participation in another investigational study that may directly or indirectly affect the results of this study within 30 days prior to the initial visit
* Allergy to the proposed anesthetic agents (e.g. nitrous oxide, midazolam, fentanyl, diphenhydramine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Intravenous sedative drug | Duration of the procedure (1-2 hours)
  Tabulate the types and dosages of intravenous sedative drugs given
Recovery time | Duration of the procedure (1-3hours)
  Time spent in procedure room to recover
Patient comfort | Duration of the procedure (1-3hours)
  Patient comfort rating intra-procedure using standardized scale
Fatigue | 24-36 hours
  The number of patients who experienced fatigue
Fatigue | 24-36 hours
  The duration of fatigue experienced, if any
Nausea/vomiting | 24-36 hours
  Number of patients who experienced nausea/vomiting
Nausea/vomiting | 24-36 hours
  Duration of nausea/vomiting
Mental Fogginess post-procedure/sedation | 24-36 hours
  Duration of mental fogginess following the procedure/sedation
Mental Fogginess post-procedure/sedation | 24-36 hours
  Number of patients who experienced mental fogginess post-procedure/sedation
Return to baseline function | 24-36 hours
  Number of hours post-procedure/sedation for patient to return to baseline function

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No